CLINICAL TRIAL: NCT00481832
Title: Autologous Followed by Non-myeloablative Allogeneic Transplantation for Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Accrual Factor
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Wen-Kai Weng, Associate Professor of Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-05730; 97623 (Other: Stanford University Alternate IRB Approval Number); BMT185 (Other: OnCore)
Record Dates: First submitted 2007-05-31; First posted 2007-06-04 (Estimated); Results first posted 2018-02-14 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-01

CONDITIONS: Lymphoma, Non-Hodgkin
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Cyclophosphamide; Carmustine; Etoposide; etoposide phosphate; Filgrastim; Granulocyte Colony-Stimulating Factor; Colony-Stimulating Factors; Antilymphocyte Serum; Cyclosporine; Mycophenolic Acid; Rituximab; Transplantation; betibeglogene autotemcel; Methylprednisolone Hemisuccinate; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- T & B Cell Mobilization Auto & Allo HCT (Experimental): A transplant regimen that conditions the subjects using total lymphoid irradiation (TLI) and anti-thymocyte globulin(ATG) which will reduce acute graft-vs-host disease to negligible rates while maintaining the anti-tumor graft vs lymphoma GvL benefit. Along with TLI/ATG regiment; Solumedrol will be used as pre-medication and anti-emetic for any side effects. For stem cell mobilization, participants will be given either B Cell NLH or T Cell NHL. Before the filgrastim (G-CSF) mobilized PBPC infusion: acetaminophen, diphenhydramine and hydrocortisone will also be given as another set of pre-medications. BCNU, Etoposide, and Cyclophosphamide will be used as a preparative regimen. Cyclosporine and mycophenolate mofetil will be administered as an immunosuppressant after transplantation. Lastly, rituximab will be infused at the end of the transplantation regimen.
  Interventions: Drug: Cyclophosphamide; Drug: BCNU; Drug: Etoposide; Drug: Filgrastim; Drug: Antithymocyte globulin; Drug: Cyclosporine; Drug: Mycophenolate mofetil; Drug: Rituximab; Procedure: Autologous hematopoietic stem cell transplantation (auto-HSCT); Procedure: Allogeneic hematopoietic stem cell transplantation (allo-HSCT); Procedure: Total lymphoid irradiation; Drug: CD34+ Cells; Drug: Solu-Medrol

INTERVENTIONS:
Drug: Cyclophosphamide — 4 gm /m² IV over 2 hours on day 8
  Other Names: Cytoxan; Neosar
Drug: BCNU — The dose of BCNU will be based on actual body weight unless the actual body weight is more than 15 kg greater than the ideal body weight in which case the adjusted ideal body weight will be used:
  Males IBW = 50 kg + 2.3 kg/inch over 5 feet Females IBW = 45.5 kg + 2.3 kg/inch over 5 feet Adjusted IBW = IBW + 50% (actual weight - IBW)
  Other Names: BiCNU; Carmustine
Drug: Etoposide — 60mg/kg, IV over 4 hours on day -4 pre-transplant and for preparative regimen. The dose of etoposide for mobilization is 2 gm/ m².
  Other Names: Eposin; Etopophos; VP-16
Drug: Filgrastim — 10µg/kg sc qd starting day following cyclosphamide (or VP-16) until last day of apheresis
  Other Names: Granulocyte colony-stimulating factor (G-CSF, GCSF); Colony-stimulating factor (CSF) 3
Drug: Antithymocyte globulin — 1.5 mg/kg/d, IV from day -11 to -7
  Other Names: ATG
Drug: Cyclosporine — 5mg/kgbid,variable, po or IV
  Other Names: cyclosporin; cyclosporin A
Drug: Mycophenolate mofetil — 15 mg/kg po on day 0, at 5-10 hours after mobilized PBPC infusion is complete. Thereafter, beginning on day +1 MMF is taken at 15 mg/kg po b.i.d. (30 mg/kg/day) if transplantation was using a matched related donor and 15 mg/kg po t.i.d if from a matched unrelated donor or a one antigen mismatched donor. Doses will be rounded up to the nearest 250 mg (capsules are 250 mg). MMF will be stopped on day +28 for matched related donors. For one antigen mismatched related or unrelated donors, the taper will begin on day +40. MMF will be tapered by 10% weekly till off, typically by day +96. If there is nausea and vomiting at any time preventing the oral administration of MMF, MMF should be administered intravenously at an equal dose. MMF dosing is based on actual body weight.
  Other Names: MMF; CellCep
Drug: Rituximab — 375 mg/m2 IV (calculated based on actual body weight) on day 1 and day 7. Administered per current standard of care..
  Other Names: Rituxan; MabThera
Procedure: Autologous hematopoietic stem cell transplantation (auto-HSCT) — Auto-HCT involves an intravenous infusion of a participant's previously collected and frozen white blood cells collected after treatment with mobilizing agents
  Other Names: Autologous peripheral blood progenitor cell (PBPC) transplantation
Procedure: Allogeneic hematopoietic stem cell transplantation (allo-HSCT) — Allo-HCT involves an intravenous infusion of a donor's white blood cells collected after treatment with mobilization with filgrastim (G-CSF)
  Other Names: Allogeneic peripheral blood progenitor cell (PBPC) transplantation
Procedure: Total lymphoid irradiation — TLI is administered in 80cGy fractions on Days -11 to Day-7 relative to allo-HSCT
  Other Names: TLI
Drug: CD34+ Cells — 2 x 10e6 CD34+ cells per kg actual body weight on Day 0
Drug: Solu-Medrol — 1 mg/kg, Day-11 to Day-7
  Other Names: Methylprednisolone

SUMMARY:
The purpose of this trial is to develop an alternative treatment for patients with poor risk non-Hodgkin's lymphoma. This trial uses a combination of high dose chemotherapy with stem cell transplant using the patient's own cells. This is followed with non-myeloablative transplant using stem cells from a related or unrelated donor to try and generate an anti-lymphoma response from the new immune system.

DETAILED DESCRIPTION:
Currently, patients with recurrent or primary refractory non-Hodgkin's lymphoma are treated with second-line chemotherapy (usually 2-3 courses) for the purpose of cytoreduction and to establish sensitivity to chemotherapy. Thereafter, peripheral blood progenitor cells are mobilized with cyclophosphamide and granulocyte colony stimulating factor, apheresed and cryopreserved. The standard high dose regimen consists of augmented carmustine, etoposide and cyclophosphamide. Unfortunately, there are subgroups of patients with poor outcomes using autologous transplantation including those with transformed lymphoma as well as patients who do not attain a minimal disease state due to chemoresistant disease.

These groups of patients have limited disease control and survival with standard chemotherapy regimens, and although they often have excellent cytoreduction with the high-dose chemotherapy regimen, relapse remains the primary cause of treatment failure. The current trial utilizes a similar approach that has been taken with patients with multiple myeloma, who appear to benefit from an allogeneic graft-versus-tumor effect, using a combined autologous and non-myeloablative allogeneic transplant regimen to reduce transplant-related complications. Eligible patients will be treated with high-dose chemotherapy using BCNU, etoposide and cyclophosphamide with autologous hematopoietic cell support as a method of cytoreduction. Approximately 60-120 days after the autologous transplant, patients will receive an allogeneic transplant using a preparative regimen of total lymphoid irradiation and anti-thymocyte globulin in an attempt to develop a graft-versus-lymphoma effect.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70 years.
* Histologically proven non-Hodgkin's lymphoma
* Relapse after achieving initial remission or failure to achieve initial remission.
* KPS > 70%
* Matched related or unrelated donor identified and available. Donor must be a complete match or have only a single allele mismatch.
* Recent Bone marrow biopsy and cytogenetic analysis
* Patients must have a pretreatment serum bilirubin < 2 x the institutional ULN, a serum creatinine < 2 x the institutional ULN and measured or estimated creatinine clearance > 50 cc/min by the following formula (all tests must be performed within 28 days prior to mobilization ): Estimated Creatinine Clearance = (140 age) X WT(kg) X 0.85 if female 72 X serum creatinine(mg/dl).
* Patients must have an EKG within 42 days prior to registration that shows no significant abnormalities that are suggestive of active cardiac disease.
* Patients must have an echocardiogram or MUGA scan within 42 days of registration. If the ejection fraction is < 40%, the patient will not be eligible. If the ejection fraction is 40-50%, patients must have an exercise echocardiogram or dobutamine-echo with a normal response to exercise.
* Patients must have a corrected diffusion capacity > 50% prior to the autologous transplant and > 40% prior to the allogeneic transplant.
* Patients with known allergy to etoposide or a history of Grade 3 hemorrhagic cystitis with cyclophosphamide are not eligible.
* Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines.

Exclusion Criteria:

* Pregnant or breast-feeding women are ineligible due to the known birth defects association with the treatments used in this study.
* Patients known to be human immunodeficiency virus (HIV)-positive are ineligible because the concern for opportunistic infection and hematologic reserve are considered to be significantly greater in this population.
* Patients with prior maligancies diagnosed > 5 years ago without evidence of disease are eligible. Patients with a prior malignancy treated < 5 years ago but have a life expectancy of > 5 years for that malignancy are eligible.
* Patients with uncontrolled infection.
* No prior autologous or allogeneic hematopoietic cell transplantation.

Donor Selection/Evaluation:

* Related or unrelated HLA identical donors who are in good health and have no contra-indication to donation.
* No contra-indication for the donor to collection by apheresis of mononuclear cells mobilized by G-CSF at a dose of 16 µg/kg of body weight.
* Virology testing including CMV, HIV, EBV, HTLV, RPR, Hepatitis A, B and C will be performed within 30 days of donation.
* No prior malignancy is allowed except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer or other cancer for which the donor has been disease-free for five years

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-01; Primary Completion 2014-10-27 (Actual); Study Completion 2017-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Kai Weng, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Enrollment
Arm/Group | T & B Cell Mobilization Auto & Allo HCT
Started | 50
Completed | 40
Not Completed | 10
Not completed — Physician Decision | 8
Not completed — Unable to collect enough stem cells | 2
Period: Autologous Hematopoietic Cell Transplant
Arm/Group | T & B Cell Mobilization Auto & Allo HCT
Started | 40
Completed | 40
Not Completed | 0
Period: Inter-transplant Period
Arm/Group | T & B Cell Mobilization Auto & Allo HCT
Started | 40
Completed | 13
Not Completed | 27
Not completed — Adverse Event | 4
Not completed — Death | 3
Not completed — Physician Decision | 4
Not completed — Disease relapse | 11
Not completed — Lack of allogeneic donor | 5
Period: Allogenic Hematopoietic Cell Transplant
Arm/Group | T & B Cell Mobilization Auto & Allo HCT
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | T & B Cell Mobilization Auto & Allo HCT
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 43
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 44
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 2
  White | 38
  More than one race | 1
  Unknown or Not Reported | 5

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival (EFS)
Description: Event-free survival (EFS) as determined for participants who receive both planned transplants, for a minimum of 3 years.
  Events are defined as "disease progression/relapse" and "death of all causes".
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | T & B Cell Mobilization Auto & Allo HCT
Number analyzed (Participants) | 13
percentage of participants | 35 [27 to 80]

2. Secondary Outcome: Incidence of Chemotherapy-associated Pneumonitis
Description: Interstitial pneumonitis (IP) is a risk associated with high-dose carmustine (BCNU) or other chemotherapy drugs used for transplantation. IP is diagnosed by 1) a decrease of >25% in DLCO compared with pre-transplant PFT DLCO values or 2) a drop of 7% or more in oxygen saturation after exertion.
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | T & B Cell Mobilization Auto & Allo HCT
Number analyzed (Participants) | 40
Participants | 16

3. Secondary Outcome: Relapse Rate
Description: Relapse rate (disease recurrence) 3 years after transplant, for participants who received both transplants, as determined by Kaplan-Meier estimation.
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | T & B Cell Mobilization Auto & Allo HCT
Number analyzed (Participants) | 13
percentage of participants | 27 [10 to 62]

4. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) 3 years after transplant, for participants who received both transplants, as determined by Kaplan-Meier estimation.
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | T & B Cell Mobilization Auto & Allo HCT
Number analyzed (Participants) | 13
percentage of participants | 57 [26 to 79]

5. Secondary Outcome: Incidence of Acute Graft Versus Host Disease (GvHD)
Description: The development of GvHD in vaccinated patients of any grade and at 6 months.
Time Frame: 6 Months
Population: Only 13 participants received both therapies and were evaluated for GVHD
Measure: Count of Participants; unit: Participants
Arm/Group | T & B Cell Mobilization Auto & Allo HCT
Number analyzed (Participants) | 13
Participants | 3

6. Secondary Outcome: Incidence of Chronic Graft Versus Host Disease (GvHD)
Description: The development of GvHD in vaccinated patients of any grade at 6 months.
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | T & B Cell Mobilization Auto & Allo HCT
Number analyzed (Participants) | 13
Participants | 3

7. Secondary Outcome: Overall Mortality Rate
Description: Overall mortality is determined by Kaplan-Meier estimation. The overall morality rate is expressed as the percentage of patients who died for any reason, including disease-related death.
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | T & B Cell Mobilization Auto & Allo HCT
Number analyzed (Participants) | 40
percentage of participants | 56 [42 to 71]

8. Secondary Outcome: Median Time to Neutrophile Engraftment
Description: Complete blood counts were measured daily after allogeneic transplant. Time to neutrophil engraftment is defined as the number of days it takes to reach an absolute neutrophils count (ANC) >500, counting from the day of transplant.
Time Frame: up to 45 days
Measure: Median (Full Range); unit: Days
Arm/Group | T & B Cell Mobilization Auto & Allo HCT
Number analyzed (Participants) | 13
Days | 17 [9 to 26]

9. Secondary Outcome: Achieving Full Donor Chimerism
Description: Achieving full donor chimerism (donor T cells >95%): Blood was sent for donor cell percentage measured by short tandem repeat (STR) at post-transplant Day 30; Day 60; Day 90; Day 120; Day 180; Day 270; and Day 360. Full donor chimerism is defined as donor CD3+ cells > 95%.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | T & B Cell Mobilization Auto & Allo HCT
Number analyzed (Participants) | 13
Participants | 10

10. Secondary Outcome: Median Time to Platelet Engraftment
Description: Complete blood counts were measured daily after allogeneic transplant. Time to platelet engraftment is defined as the number of days it takes to reach platelet count >20,000, counting from the day of transplant.
Time Frame: Up to 45 days
Measure: Median (Full Range); unit: Days
Arm/Group | T & B Cell Mobilization Auto & Allo HCT
Number analyzed (Participants) | 13
Days | 11 [1 to 41]

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | T & B Cell Mobilization Auto & Allo HCT
All-Cause Mortality (participants affected / at risk) | 24/50
Serious Adverse Events (participants affected / at risk) | 5/50
Other Adverse Events (participants affected / at risk) | 4/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T & B Cell Mobilization Auto & Allo HCT (N=50)
Viral Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Adult Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal/ Liver failure (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T & B Cell Mobilization Auto & Allo HCT (N=50)
Decreased platelet count (Blood and lymphatic system disorders) | 2 (2)
Decreased lung persusion capacity (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Decreased neutrophile count (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No